CLINICAL TRIAL: NCT04876950
Title: Post Discharge After Surgery Virtual Care with Remote Automated Monitoring Technology-2 (PVC-RAM-2) Trial
Acronym: PVC-RAM-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1.0.2021.04.30
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Surgery; Perioperative Complication
Keywords: Virtual care; Remote monitoring; Acute hospital care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Care with Remote Automated Monitoring (Experimental): Patients randomized to the PVC-RAM-2 intervention will take biophysical measurements with the RAM technology and complete a daily recovery survey for 14 days after index hospital discharge, and nurses will review these results daily. Through scheduled video visits, patients will virtually interact with a nurse on days 1, 3, 7 and 14, and a physician on days 1 and 14. Patients will take a photograph of their wound daily for the first 7 days on the program, and nurses will review these pictures. If the patient's RAM measurements exceed predetermined thresholds, the patient reports specific symptoms (e.g., shortness of breath), a drug error is identified, or the virtual nurse has concerns about the patient's health that they cannot resolve, they will escalate care to a pre-assigned and available physician. Two 7-day extensions to the intervention will be possible, based on the patient's need for continued support. This decision will be based on standardized criteria.
  Interventions: Combination Product: Virtual care with remote automated monitoring
- Standard Care (No Intervention): Patients randomized to standard care will receive post discharge care as per the standard of care at the hospital where they undergo surgery.

INTERVENTIONS:
Combination Product: Virtual care with remote automated monitoring — Use of Cloud Diagnostics connected health kit for at home monitoring with virtual clinical from nursing and perioperative physician team.
  Arms: Virtual Care with Remote Automated Monitoring

SUMMARY:
The Post discharge after surgery Virtual Care with Remote Automated Monitoring technology-2 (PVC-RAM-2) Trial is a multicentre, parallel group, superiority, randomized controlled trial to determine the effect of virtual care with remote automated monitoring (RAM) technology compared to standard care on acute-hospital care during the 45-day follow up after randomization, in adults who have undergone semi-urgent (e.g., oncology), urgent (e.g., hip fracture), or emergency (e.g., ruptured abdominal aortic aneurysm) surgery. Secondary outcomes at 45 days after randomization include 1) days in hospital; 2) index length of hospital stay; 3) hospital re-admission; 4) emergency department visit; 5) medication error detection; 6) medication error correction; and 7) surgical site infection. Additional secondary outcomes are pain of any severity, and moderate-to-severe pain assessed at 15 and 45 days. We will also assess optimal management of long-term health by evaluating among self-reported current smokers and those with atherosclerotic disease, whether patients are taking classes of efficacious medications at 45 days post randomization.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥40 years of age;
2. will undergo or have undergone semi-urgent, urgent, or emergency surgery requiring expected hospital stay of ≥2 days; and
3. provide informed consent to participate.

Exclusion Criteria:

1. planned transfer to a rehabilitation or convalescent facility, or repatriation from trial hospital site to local community hospital following surgery;
2. are unable to communicate with research staff, complete study surveys, or undertake an interview using a tablet computer due to a language barrier or a cognitive, visual, or hearing impairment; or
3. reside in an area without cellular network coverage.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acute-hospital care | 45 days post randomization
  Composite outcome of hospital re-admission and emergency department visit, which includes urgent-care centre visit.

SECONDARY OUTCOMES:
Days in hospital | 45 days post randomization
  Total number of days in hospital from randomization to 45 days post-randomization, including index hospital stay and any hospital readmission (s). A day in hospital is counted if a participant spends 1 minute of any day admitted to hospital.
Index length of hospital stay | 45 days post randomization
  Length of hospital stay calculated from time of surgery completion (i.e., time of surgical wound closure) until discharge from the index hospitalization (measured in days and hours).
Hospital readmission | 45 days post randomization
  Patient admission to an acute-care hospital.
Emergency department visit | 45 days post randomization
  Patient visit to an emergency department.
Medication error detection | 45 days post randomization
  Medication errors include mistakes in medication prescribing, transcribing, dispensing, administering, or monitoring due to preventable events or actions taken by a patient, caregiver, or healthcare worker. Medication errors include: drug omission (i.e., patient did not take a drug they were supposed to take), drug commission (i.e., patient taking a drug they were not supposed to take), duration error, dosing error, frequency error, route error, and timing error. We will record all drug errors identified and also report whether they resulted in harm.
Medication error correction | 45 days post randomization
  Any medication error that is corrected.
Surgical site infection | 45 days post randomization
  Surgical site infection is an infection that occurs within 30 days after randomization and involves the skin, subcutaneous tissue of the incision (superficial incisional), or the deep soft tissue (e.g., fascia, muscle) of the incision (deep incisional).
Pain of any severity | 15 and 45 days post randomization
  Pain intensity and related interference with usual daily activities, will be measured via the Brief Pain Inventory-Short Form (BPI-SF).The BPI-SF includes four 11-point numeric rating scales (NRS) of pain intensity, which measure "average", "least", and "worst" pain intensity in the past 24 hours (hrs.), respectively, as well as pain intensity "now" (0= no pain, 10= pain as bad as you can imagine).
Moderate to severe pain | 15 and 45 days post randomization
  Pain intensity and related interference with usual daily activities, will be measured via the Brief Pain Inventory-Short Form (BPI-SF).The BPI-SF includes four 11-point numeric rating scales (NRS) of pain intensity, which measure "average", "least", and "worst" pain intensity in the past 24 hours (hrs.), respectively, as well as pain intensity "now" (0= no pain, 10= pain as bad as you can imagine). Pain is of moderate or greater severity is defined by a score of ≥4/10 on a standard numeric rating scale (NRS) for pain.
Optimal pharmacological management for patients with atherosclerotic disease | 45 days post randomization
  Among patients with atherosclerotic disease, we will also assess optimal pharmacological management based upon whether patients are taking 0, 1, 2, or 3 of the following classes of efficacious medications at 45 days (i.e., an antiplatelet or anticoagulant drug; an angiotensin-converting enzyme inhibitor or angiotensin-receptor blocker; and a statin).
Optimal pharmacological management self-reported current smokers | 45 days post randomization
  Among patient who self-report to be current smokers at baseline, we will assess if patients are receiving pharmacological smoking cessation interventions at 45 days after randomization.

OTHER OUTCOMES:
Infection | 45 days post randomization
  Infection is defined as a pathologic process caused by the invasion of normally sterile tissue, fluid, or body cavity by pathogenic or potentially pathogenic organisms.
Re-operation | 45 days post randomization
  Re-operation refers to any surgical procedure undertaken for any reason (e.g., wound dehiscence, infection).
Myocardial Infarction | 45 days post randomization
  4th Universal definition of myocardial infarction.
Acute Heart Failure | 45 days post randomization
  The definition of acute heart failure requires at least one of the following clinical signs (i.e., elevated jugular venous pressure, respiratory rales or crackles, crepitations, or presence of S3) with at least one of the following:
  1. radiographic findings of vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema, OR
  2. heart failure treatment with a diuretic and documented clinical improvement.
Arrhythmia that results in patient presenting to an emergency department or being admitted to hospital | 45 days post randomization
  Any arrhythmia that results in patient presenting to an emergency department, which includes an urgent care centre, or being admitted to hospital.
Death | 30 days post randomization
  All cause mortality.
Health-related quality of life (HRQL) | 45 days post randomization
  HRQL will be measured with the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) instrument (https://euroqol.org/eq-5d-instruments/sample-demo) due to its increased sensitivity and validation in several countries including Canada. The EQ-5D-5L is also recommended in Canada to calculate the Quality Adjusted Life Years (QALYs) when conducting cost-effectiveness analyses.
  The EQ-5D-5L questionnaire consists of descriptive questions regarding 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with a 5-level scale for participants to indicate the most accurate response (ranging from no problems to extreme problems).
Health services utilization-related costs | 45 days post randomization
  Costs associated with hospital re-admission, length of stay, and healthcare utilization will be obtained from administrative datasets.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGillion, PhD, Principal Investigator — McMaster University, Population Health Research Institute; PJ Devereaux, M.D, PhD, Principal Investigator — McMaster University, Population Health Research Institute; Sandra Ofori, M.D., PhD, Principal Investigator — Hamilton Health Sciences, Population Health Research Institute
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No